CLINICAL TRIAL: NCT06313762
Title: Use of Virtual Reality in the Reduction of Pain After the Administration of Vaccines Among Children in Primary Care Centers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Mercedes de la Cruz Herrera, Principal Investigator, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Codi CEIm: 21/132-P
Record Dates: First submitted 2024-02-22; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Pain; Pediatrics; Vaccination; Virtual Reality
MeSH Terms: conditions — Pain | interventions — Aging; Hepatitis A Vaccines

STUDY DESIGN:
Intervention Model Description: The intervention group will use the Pico G2 VR goggles (Pico Interactive Inc) during the administration of the two vaccines, together with an Android AOYODKG tablet, which will be connected to the goggles as a controller.
  The control group participants will receive traditional distractors, such as being held by the parent or guardian who accompanies them to the appointment, receiving stickers at the end of the appointment, or receiving rewards that the parent or guardian has prepared from home.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Device: Pico G2 Virtual Reality Glasses (Pico Interactive Inc), together with an Android AOYODKG tablet; Biological: Triple Viral + Varicella Vaccine at 3 years of age; Biological: Hepatitis A + Diphtheria-Tetanus-Pertussis Vaccine at 6 years of age.
- Control Group (Active Comparator)
  Interventions: Behavioral: Traditional Distractors; Biological: Triple Viral + Varicella Vaccine at 3 years of age; Biological: Hepatitis A + Diphtheria-Tetanus-Pertussis Vaccine at 6 years of age.

INTERVENTIONS:
Device: Pico G2 Virtual Reality Glasses (Pico Interactive Inc), together with an Android AOYODKG tablet — They will experience in first person the two and a half minute graphic adventure, called Leia&amp;#39;s World, during the administration of the vaccines.
  Arms: Intervention Group
Behavioral: Traditional Distractors — The control group participants will receive traditional distractors, such as being held by the parent or guardian who accompanies them to the appointment, receiving stickers at the end of the appointment, or receiving rewards that the parent or guardian has prepared from home, during the administration of the vaccines.
  Arms: Control Group
Biological: Triple Viral + Varicella Vaccine at 3 years of age — Administration of vaccines in 3-year-old children, as appropriate according to the vaccination schedule
Biological: Hepatitis A + Diphtheria-Tetanus-Pertussis Vaccine at 6 years of age. — Administration of vaccines in 6-year-old children, as appropriate according to the vaccination schedule.

SUMMARY:
The objective of this randomized, multicenter, open-label, parallel, controlled clinical trial is to evaluate pain reduction during the administration of two vaccines in children aged 3 and 6 years through virtual reality.

The main question[s] it aims to answer are:

1. To evaluate the reduction in pain during the administration of two vaccines in children aged 3 and 6 years.
2. To evaluate the reduction in anxiety during and after the administration of two vaccines in children aged 3 and 6 years.
3. Improve the satisfaction of parents or legal guardians after the administration of two vaccines in children aged 3 and 6 years.
4. Evaluate the Safety of the use of virtual reality glasses in children aged 3 and 6 years during the administration of vaccines.

The study population will include children aged 3 and 6 years who are included in the patient registry and are being seen in a primary care center of the Catalan Institute of Health in Central Catalonia.

The clinical trial has two assigned groups: a control group and an intervention group.

The intervention group will use the Pico G2 VR goggles (Pico Interactive Inc) during the administration of the two vaccines, together with an Android AOYODKG tablet, which will be connected to the goggles as a controller.

The control group participants will receive traditional distractors, such as being held by the parent or guardian who accompanies them to the appointment, receiving stickers at the end of the appointment, or receiving rewards that the parent or guardian has prepared from home.

International Registered Report Identifier (IRRID): PRR1-10.2196/35910

DETAILED DESCRIPTION:
The participants will be selected from a patient diary register. Both the sequence and the allocation of participants to the interventions will be generated by using the RandomizedR computer system.

Due to the nature of the study, it will not be possible to mask patients or health care professionals. Therefore, the trial will be open or unblinded. However, a blind evaluation by third parties will be carried out, as the person in charge of data analysis will not be involved with the intervention.

To detect a 1-point difference between the two groups on the pain level scale, a sample of 150 boys and girls in each group is required, assuming an SD of 3 points, an α risk of 5%, a power of 80%, and an estimated loss to follow-up rate of 5%.

The data will be obtained through Microsoft Forms (anapplication included in Office 365 [Microsoft Corporation] that allows one to create customized questionnaires, surveys, and records) and analyzed with R software (version 4.0.3).

ELIGIBILITY:
Inclusion Criteria:

The patients who will take part in the study will be those from the pediatric population (ie, those aged 3 and 6 years) in the register of patients from a primary care center of the Catalan Institute of Health in Central Catalonia who, according to the vaccination schedule, are due to receive 1 of the following 2 vaccinations:

1. the triple viral+varicella vaccine at 3 years of age.
2. the hepatitis A+diphtheria-tetanus-pertussis vaccine at age 6.

Exclusion Criteria:

1. Patients who have already received 1 of the 2 vaccines to be administered.
2. Patients and accompanying persons who do not understand and speak Catalan or Spanish.
3. Patients with physical or mental illnesses, as well as those with blindness or deafness.
4. Patients with a known history of epileptic episodes or severe motion sickness.
5. Patients with autism spectrum disorder.
6. patients with any infections, burns, or injuries to the face, head, or neck that may interfere with the placement of the VR device.
7. the absence of legal guardians for signing the informed consent form.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain perception during the administration of two vaccines in children aged 3 and 6 years, through the Wong-Baker Pain Scale. | Up to 24 months
  O: no hurt, 2: hurts little bit, 4: hurts little more, 6: hurts even more, 8: hurts whole lot, 10: hurts worst

SECONDARY OUTCOMES:
Evaluation of anxiety during the administration of two vaccines in children aged 3 and 6 years, through heart rate and the Children's Fear Scale. | Up to 24 months
  0: no anxiety, 1: mild anxiety, 2: moderate anxiety, 3: severe anxiety, 4: very severe anxiety
Degree of satisfaction of parents/legal guardians of minors after the administration of two vaccines, using the CSAT scale. | Up to 24 months
  Not at all satisfied, slightly satisfied, normal, satisfied, very satisfied.
Number of patients who experienced adverse effects during the administration of vaccines and who used virtual reality glasses, through the registration of the effects presented. | Up to 24 months
  Record of adverse effects: None, fall, seizures, loss of consciousness, blurred vision, dizziness, nausea, headache, others.

CONTACTS AND LOCATIONS:
Locations (1):
- Catalan Institute of Health. Territorial Management of Central Catalonia., Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De La Cruz Herrera M, Fuster-Casanovas A, Miro Catalina Q, Cigarrran Mensa M, Vilanova Guitart I, Aguera Sedeno A, Vidal-Alaball J, Grau Carrion S. Use of virtual reality in the reduction of pain after the administration of vaccines among children in primary care centers in Central Catalonia: Randomized clinical trial. PLoS One. 2025 May 7;20(5):e0322840. doi: 10.1371/journal.pone.0322840. eCollection 2025. PMID 40334011
- See also: Protocol: Use of Virtual Reality in the Reduction of Pain After the Administration of Vaccines Among Children in Primary Care Centers: Protocol for a Randomized Clinical Trial. — https://www.researchprotocols.org/2022/4/e35910
- Available data/document: Study Protocol: (IRRID): PRR1-10.2196/35910 — https://www.researchprotocols.org/2022/4/e35910 — Protocol: Use of Virtual Reality in the Reduction of Pain After the Administration of Vaccines Among Children in Primary Care Centers: Protocol for a Randomized Clinical Trial